CLINICAL TRIAL: NCT00764348
Title: Evaluation of Wound Biofilm in Acute and Chronic Wounds
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn as MSU approval obained
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-002
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Wounds
Keywords: Acute and Chronic Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — traumatic, diabetic foot ulcer, decubitus ulcer, venous leg ulcer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment
  Interventions: Other: no treatment

INTERVENTIONS:
Other: no treatment

SUMMARY:
Patients who present to a wound care center for management of their wounds will be evaluated clinically to establish if their wounds are chronic or acute. These patients will undergo standard of care management of their wounds. If debridement is indicated for the patient, the patient will be asked to participate in a study. Once the standard of care debridement is complete, the material debrided from the wound, instead of being discarded into a biohazard bag, will be prepared for shipment. The samples will then be shipped to the Center for Biofilm Engineering where microscopic evaluation will be conducted on the material. Conclusion will be made from that analysis.

DETAILED DESCRIPTION:
A planktonic concept of the bacteria present on the surface of a chronic wound is no longer viable. Microscopic studies show that biofilm is present on chronic wounds yet does not seem to be prominent on the surface of acute wounds. Biofilm is able to neutralize our host defenses and commandeer host systems, and possesses an impressive array of defenses and virulence factors. Clinically we see a significant difference in the healing behavior between chronic and acute wounds. Also, suppression of biofilm using multiple simultaneous strategies including debridement, anti-biofilm agents, specific biocides, antibiotics and advanced technologies improves wound healing. This suggests biofilm plays an important role in delayed wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute and Chronic Wounds
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
It is important for all wound care providers to firmly grasp the wound biofilm concept, its importance in delayed wound healing, and how it differs from a planktonic bacterial concept.